CLINICAL TRIAL: NCT04096274
Title: Randomized Trial of a Leadership and Organizational Change Strategy to Improve the Implementation and Sustainment of Digital Measurement-based Care in Youth Mental Health Services
Brief Title: Working to Implement and Sustain Digital Outcome Measures
Acronym: WISDOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boise State University (Other)
Collaborators: University of California, San Diego (Other); University of Central Florida (Other); University of Pennsylvania (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 8424; R01MH119127 (NIH)
Record Dates: First submitted 2019-09-09; First posted 2019-09-19 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2022-07

CONDITIONS: Implementation; Behavioral Symptoms
Keywords: LOCI; measurement-based care; evidence-based practice; behavioral health; youth mental health; leadership; implementation science
MeSH Terms: conditions — Behavioral Symptoms | interventions — Leadership

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Clinicians and caregivers of youth were naïve to condition; however, masking of clinic leaders was not possible due to the nature of the LOCI strategy (which entails leadership training and consultation).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOCI (Intervention) (Experimental): In clinics assigned to the LOCI condition, executives and first-level leaders will receive leadership training and coaching to support implementation of the OQ-A system. In addition, leaders and clinicians in this condition will receive training and technical assistance to implement the OQ-A measurement-based care system.
  Interventions: Behavioral: Leadership for Organization Change and Implementation (LOCI); Behavioral: Training and Technical Assistance Only
- Training and Technical Assistance only (Control) (Active Comparator): In clinics assigned to the control group, leaders and clinicians will receive training and technical assistance to implement the OQ-A measurement-based care system. In addition, to support enrollment in this condition, leaders in this condition will be offered access to general web-based leadership seminars.
  Interventions: Behavioral: Training and Technical Assistance Only

INTERVENTIONS:
Behavioral: Leadership for Organization Change and Implementation (LOCI) — LOCI is a multicomponent implementation strategy that engages organizational executives and first-level leaders (i.e., those who administratively supervise clinicians) to build an organizational climate to support the implementation of a focal evidence-based practice (EBP) with fidelity. In this study, the focal EBP is the OQ-A system. LOCI includes two overarching components: (1) monthly organizational strategy meetings between executives and LOCI consultants/trainers to develop and embed policies, procedures, and practices that support implementation of a focal EBP, and (2) training and coaching for first-level leaders, to develop their skills in leading implementation. The aim of these components is to develop an organizational implementation climate in which clinicians' perceive that use of the OQ-A with high fidelity is expected, supported, and rewarded.
  Arms: LOCI (Intervention)
Behavioral: Training and Technical Assistance Only — All leaders and clinicians in participating clinics will receive standardized OQ-A training and technical assistance provided by the OQ-A purveyor organization. This includes an initial, 6-hr, in-person OQ-A training; two, live, virtual, 1-hr booster trainings, offered 3 and 5 months after the initial training; and, year-round technical assistance from the OQ-A purveyor organization. Technical assistance includes virtual training sessions, online library of training videos, and customer care representative for technical support.
  In addition, to encourage participation in the study, a set of four 1-hr, web-based general leadership seminars will be offered to leaders in the control condition. These will cover topics ranging from effective leadership, to giving effective feedback.

SUMMARY:
This study will investigate the effects of an organizational implementation strategy called Leadership and Organizational Change for Implementation (LOCI), relative to training and technical assistance only, on fidelity to, and youth service outcomes of, a well-established digital measurement-based care intervention called the Outcomes Questionnaire-Analyst in outpatient community mental health clinics.

DETAILED DESCRIPTION:
Using a cluster randomized, controlled, hybrid type III effectiveness-implementation design, this trial will investigate the effects of LOCI on the fidelity and and clinical outcomes of a digital measurement-based care (MBC) system called the Outcomes Questionnaire Analyst (OQ-A). The trial will enroll up to 22 outpatient mental health clinics that serve youth and randomly assign them using covariate constrained randomization to either LOCI or training and technical assistance only. Within each clinic, up to 2 first level leaders will be recruited (max N of 40 total) and a minimum of 3 clinicians will be recruited per site (60 total). Data on youth outpatients who receive services will be collected in two phases. In each phase, a unique cohort of 360 caregivers of youth who participate in services will be sampled from the participating clinics. Caregivers will report on the service outcomes and experiences of eligible youth who receive services. The total caregiver enrollment for two phases will be 720 (360*2).

ELIGIBILITY:
Participants for this project will fall into four groups: 1) clinic executives and upper leaders (i.e., Chief Executive Officer, Executive Directors, program administrators, n=20), 2) clinic first-level leaders (i.e. clinical supervisors, n=20), 3) clinicians serving children with emotional and behavioral disorders (n=120), and 4) caregivers of children with emotional and behavioral disorders who receive outpatient mental health services within participating clinics (n=720). Caregivers will be recruited in two distinct cohorts of 360 each.

Inclusion criteria for all groups of participants are intentionally broad in line with the pragmatic nature of the trial.

Inclusion Criteria for Clinics

1. Provide outpatient psychotherapy services to children ages 4 to 18 who have emotional and/ or behavioral disorders and their families
2. Have at least 3 full time equivalent clinicians on staff
3. Not currently implementing a digital measurement-based care system clinic wide

Inclusion Criteria for Executives and Upper Leaders

1. Identified as Chief Executive Officer, Executive Director, or high-level administrator at an enrolled clinic

Inclusion Criteria for first-level leaders

1. Identified as a clinical supervisor or clinical work-group supervisor/ leader at an enrolled clinic

Inclusion Criteria for Clinicians

1. Employed as staff at participating clinic
2. Provides outpatient mental health services (psychotherapy) to youth clients

Inclusion Criteria for Caregivers of Youth Who Receive Services at Participating Clinics

1. Child is ages 4 to 18 years at intake,
2. Child has been diagnosed with an emotional or behavioral disorder by clinic staff
3. Clinical staff at the site determined that the youth's treatment needs can be appropriately addressed by the clinic

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 686 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nate Williams, PhD, Principal Investigator — Boise State University
Locations (4):
- United States (4):
  - University of California, San Diego, San Diego, California
  - University of Central Florida, Orlando, Florida
  - Boise State University, Boise, Idaho
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams NJ, Choy-Brown M, Vega N, Aarons GA, Ehrhart MG, Marcus SC. Testing normalization process theory in a randomized trial of mental health clinics implementing digital measurement-based care. Implement Sci. 2026 Feb 9. doi: 10.1186/s13012-026-01485-4. Online ahead of print. PMID 41656239
- [Derived] Williams NJ, Ehrhart MG, Aarons GA, Esp S, Sklar M, Carandang K, Vega NR, Brookman-Frazee L, Marcus SC. Improving measurement-based care implementation in youth mental health through organizational leadership and climate: a mechanistic analysis within a randomized trial. Implement Sci. 2024 Mar 28;19(1):29. doi: 10.1186/s13012-024-01356-w. PMID 38549122
- [Derived] Williams NJ, Marcus SC, Ehrhart MG, Sklar M, Esp SM, Carandang K, Vega N, Gomes AE, Brookman-Frazee L, Aarons GA. Randomized Trial of an Organizational Implementation Strategy to Improve Measurement-Based Care Fidelity and Youth Outcomes in Community Mental Health. J Am Acad Child Adolesc Psychiatry. 2024 Oct;63(10):991-1004. doi: 10.1016/j.jaac.2023.11.010. Epub 2023 Dec 7. PMID 38070868
- [Derived] Choy-Brown M, Williams NJ, Ramirez N, Esp S. Psychometric evaluation of a pragmatic measure of clinical supervision as an implementation strategy. Implement Sci Commun. 2023 Apr 6;4(1):39. doi: 10.1186/s43058-023-00419-1. PMID 37024945
- See also: Information about Leadership for Organizational Change for Implementation (LOCI). — https://www.implementationleadership.com/
- See also: Information about the digital measurement-based care system, OQ-A. — http://www.oqmeasures.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data were only collected from caregivers of youth who received services at participating clinics. Caregivers reported on youth's mental health service experiences and outcomes. Consequently, started and completed numbers shown below only reflect caregivers of eligible youth who participated in services (i.e., number of caregivers enrolled). Youths were not enrolled.
Units Other Than Participants: Clinics
Groups:
- LOCI (Intervention): In clinics assigned to the LOCI condition, executives and first-level leaders will receive leadership training and coaching to support implementation of the OQ-A system. In addition, leaders and clinicians in this condition will receive training and technical assistance to implement the OQ-A measurement-based care system.
  Leadership for Organization Change and Implementation (LOCI) is a multicomponent implementation strategy that engages organizational executives and first-level leaders (i.e., those who administratively supervise clinicians) to build an organizational climate to support the implementation of a focal evidence-based practice (EBP) with fidelity. In this study, the focal EBP is the OQ-A system. LOCI includes two overarching components: (1) monthly organizational strategy meetings between executives and LOCI consultants/trainers to develop and embed policies, procedures, and practices that support implementation of a focal EBP, and (2) training and coaching for first-level leaders, to develop their skills in leading implementation. The aim of these components is to develop an organizational implementation climate in which clinicians' perceive that use of the OQ-A with high fidelity is expected, supported, and rewarded.
  Training and Technical Assistance: All leaders and clinicians in participating clinics will receive standardized OQ-A training and technical assistance provided by the OQ-A purveyor organization.
- Training and Technical Assistance Only (Control): In clinics assigned to the control group, leaders and clinicians will receive training and technical assistance to implement the OQ-A measurement-based care system. In addition, to support enrollment in this condition, leaders in this condition will be offered access to general web-based leadership seminars.
  Training and Technical Assistance Only: All leaders and clinicians in participating clinics will receive standardized OQ-A training and technical assistance provided by the OQ-A purveyor organization. This includes an initial, 6-hr, in-person OQ-A training; two, live, virtual, 1-hr booster trainings, offered 3 and 5 months after the initial training; and, year-round technical assistance from the OQ-A purveyor organization. Technical assistance includes virtual training sessions, online library of training videos, and customer care representative for technical support.
  In addition, to encourage participation in the study, a set of four 1-hr, web-based general leadership seminars will be offered to leaders in the control condition. These will cover topics ranging from effective leadership, to giving effective feedback.
Period: Phase I
Arm/Group | LOCI (Intervention) | Training and Technical Assistance Only (Control)
Started | 117; 11 Clinics | 117; 10 Clinics
Completed | 112; 10 Clinics | 112; 8 Clinics
Not Completed | 5; 1 Clinics | 5; 2 Clinics
Not completed — Lost to Follow-up | 5 | 5
Period: Phase II
Arm/Group | LOCI (Intervention) | Training and Technical Assistance Only (Control)
Started | 269; 11 Clinics | 183; 8 Clinics
Completed | 258; 10 Clinics | 172; 8 Clinics
Not Completed | 11; 1 Clinics | 11; 0 Clinics
Not completed — Lost to Follow-up | 11 | 11

BASELINE CHARACTERISTICS:
Population: The data presented below reflects characteristics of youth as reported by their enrolled caregivers. With the exception of the family variables noted below, data on caregivers was not reported. Required fields for age, race, and sex refer to caregivers and therefore have values of 0 because this data was not reported. Please also note that the baseline characteristics shown below are reported separately for Phase I and Phase II of the trial because each phase was enrolled as a separate cohort.
Groups:
- LOCI (Intervention): The Leadership for Organization Change and Implementation (LOCI) strategy is a multicomponent implementation strategy that engages organizational executives and first-level leaders (i.e., those who administratively supervise clinicians) to build an organizational climate to support the implementation of a focal evidence-based practice (EBP) with fidelity. In this study, the focal EBP is the OQ-A system. LOCI includes two overarching components: (1) monthly organizational strategy meetings between executives and LOCI consultants/trainers to develop and embed policies, procedures, and practices that support implementation of a focal EBP, and (2) training and coaching for first-level leaders, to develop their skills in leading implementation. The aim of these components is to develop an organizational implementation climate in which clinicians' perceive that use of the OQ-A with high fidelity is expected, supported, and rewarded.
- Training and Technical Assistance Only (Control): All leaders and clinicians in participating clinics will receive standardized OQ-A training and technical assistance provided by the OQ-A purveyor organization. This includes an initial, 6-hr, in-person OQ-A training; two, live, virtual, 1-hr booster trainings, offered 3 and 5 months after the initial training; and, year-round technical assistance from the OQ-A purveyor organization. Technical assistance includes virtual training sessions, online library of training videos, and customer care representative for technical support.
  In addition, to encourage participation in the study, a set of four 1-hr, web-based general leadership seminars will be offered to leaders in the control condition. These will cover topics ranging from effective leadership, to giving effective feedback.
- Total: Total of all reporting groups
Arm/Group | LOCI (Intervention) | Training and Technical Assistance Only (Control) | Total
Number analyzed (Participants) | 386 | 300 | 686
Age, Categorical [Count of Participants; unit: Participants] — Population: Data not collected from caregivers for this baseline measure
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Data not collected from caregivers for this baseline measure
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data not collected from caregivers for this baseline measure
Phase I: Youth Short-form Assessment for Children (SAC) Total Problem Score [Mean (Standard Deviation); unit: units on a scale] — The SAC Total Problem Score is a 48-item measure of youth internalizing (e.g., anxious, depressed) and externalizing (e.g., aggressive, noncompliant, overactive) behaviors (range=0-96). It has extensive evidence of score reliability and validity in clinical and non-clinical samples as well as sensitivity to change in randomized trials. Higher scores indicate more problems. The clinical cut score is 26. Population: Data for Phase I only
  units on a scale
    number analyzed (Participants) | 117 | 117 | 234
    (all) | 37.1 (13.6) | 34.1 (12.8) | 35.6 (13.2)
Phase I: Youth received prior mental health treatment [Count of Participants; unit: Participants] — Population: Data for Phase I only
  Participants
    number analyzed (Participants) | 117 | 117 | 234
    (all) | 66 | 58 | 124
Phase I: Family Income [Count of Participants; unit: Participants] — Population: Data for Phase I only
  Participants
    number analyzed (Participants) | 117 | 117 | 234
    Less than $25,750 | 27 | 20 | 47
    $25,751 to $35,535 | 19 | 18 | 37
    $35,536 to $51,500 | 19 | 20 | 39
    More than $51,500 | 50 | 59 | 109
    Unknown or not reported | 2 | 0 | 2
Phase I: Parent Highest Education Level [Count of Participants; unit: Participants] — Population: Data for Phase I only
  Participants
    number analyzed (Participants) | 117 | 117 | 234
    High school graduate/GED or less | 25 | 23 | 48
    Associate's degree or some college | 48 | 42 | 90
    Bachelor's degree | 26 | 28 | 54
    Graduate degree | 18 | 24 | 42
    Unknown or not reported | 0 | 0 | 0
Phase I: Youth age [Mean (Standard Deviation); unit: years] — Population: Data for Phase I only
  years
    number analyzed (Participants) | 117 | 117 | 234
    (all) | 11.3 (3.7) | 12.1 (4.0) | 11.7 (3.8)
Phase I: Youth sex [Count of Participants; unit: Participants] — Population: Data for Phase I only
  Participants
    number analyzed (Participants) | 117 | 117 | 234
    Male | 54 | 54 | 108
    Female | 62 | 63 | 125
    Prefer not to disclose | 1 | 0 | 1
Phase I: Youth Race [Count of Participants; unit: Participants] — Population: Data for Phase I only
  Participants
    American Indian or Alaskan Native: number analyzed (Participants) | 117 | 117 | 234
    American Indian or Alaskan Native | 1 | 2 | 3
    Asian | 1 | 1 | 2
    Black or African American | 1 | 2 | 3
    Multiracial | 10 | 6 | 16
    Pacific Islander or Hawaiian Native | 0 | 0 | 0
    Prefer to self-describe | 3 | 2 | 5
    White | 98 | 103 | 201
    Prefer not to disclose | 3 | 1 | 4
Phase I: Youth Hispanic/ Latinx Ethnicity [Count of Participants; unit: Participants] — Population: Date for Phase I only
  Participants
    number analyzed (Participants) | 117 | 117 | 234
    (all) | 21 | 14 | 35
Phase II: Youth Short-form Assessment for Children (SAC) Total Problem Score [Mean (Standard Deviation); unit: units on a scale] — The SAC Total Problem Score is a 48-item measure of youth internalizing and externalizing behaviors (range=0-96). It has extensive evidence of score reliability and validity in clinical and non-clinical samples as well as sensitivity to change in randomized trials. Higher scores indicate more problems. The clinical cut score is 26. Population: Data for Phase II only
  units on a scale
    number analyzed (Participants) | 269 | 183 | 452
    (all) | 35.1 (13.3) | 34.7 (13.6) | 34.9 (13.4)
Phase II: Youth received prior mental health treatment [Count of Participants; unit: Participants] — Population: Data for Phase II only
  Participants
    number analyzed (Participants) | 269 | 183 | 452
    (all) | 153 | 110 | 263
Phase II: Family income [Count of Participants; unit: Participants] — Population: Data for Phase II only
  Participants
    number analyzed (Participants) | 269 | 183 | 452
    Less than $25,750 | 57 | 34 | 91
    $25,751 to $35,535 | 45 | 25 | 70
    $35,536 to $51,500 | 55 | 29 | 84
    More than $51,500 | 107 | 91 | 198
    Unknown | 5 | 4 | 9
Phase II: Parent Highest Education Level [Count of Participants; unit: Participants] — Population: Data for Phase II only
  Participants
    number analyzed (Participants) | 269 | 183 | 452
    High school graduate/ GED or less | 37 | 29 | 66
    Associate's degree or some college | 129 | 76 | 205
    Bachelor's degree | 64 | 53 | 117
    Graduate degree | 34 | 25 | 59
    Unknown | 5 | 0 | 5
Phase II: Youth age [Mean (Standard Deviation); unit: years] — Population: Data for Phase II only
  years
    number analyzed (Participants) | 269 | 183 | 452
    (all) | 10.5 (3.6) | 11.6 (3.8) | 10.9 (3.7)
Phase II: Youth sex [Count of Participants; unit: Participants] — Population: Data for Phase II only
  Participants
    number analyzed (Participants) | 269 | 183 | 452
    Male | 118 | 67 | 185
    Female | 149 | 114 | 263
    Prefer not to disclose | 2 | 2 | 4
Phase II: Youth race [Count of Participants; unit: Participants] — Population: Data for Phase II only
  Participants
    number analyzed (Participants) | 269 | 183 | 452
    American Indian or Alaskan Native | 5 | 0 | 5
    Asian | 3 | 2 | 5
    Black or African American | 2 | 3 | 5
    Pacific Islander or Hawaiian Native | 1 | 0 | 1
    Prefer not to disclose | 3 | 0 | 3
    Prefer to self-describe | 12 | 5 | 17
    Multiracial | 20 | 13 | 33
    White | 223 | 160 | 383
Phase II: Youth Hispanic/ Latinx Ethnicity [Count of Participants; unit: Participants] — Population: Data for Phase II only
  Participants
    number analyzed (Participants) | 269 | 183 | 452
    (all) | 40 | 21 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage Fidelity to the OQ-A System Experienced by the Youth (0-100%)
Description: Fidelity to the OQ-A will be measured by using electronic meta-data from the OQ-A system combined with caregiver reported information on the number of sessions the youth attended. For each youth, a fidelity index will be generated that represents the product of two quantities: (a) the youth's completion rate (i.e., number of measures administered relative to the number of sessions attended within the 6-month observation period), and (b) the youth's viewing rate (i.e., the number of feedback reports viewed by the clinician relative to the number of measures administered). Note that this product is equivalent to the ratio of viewed feedback reports to total sessions; it represents an events/trials proportion. MBC fidelity index scores summarize the level of MBC fidelity experienced by each youth (range=0-1). Higher scores indicate the youth experienced greater fidelity to MBC.
Time Frame: 0-6 months after youth's baseline/ entry into treatment
Population: Youths from the Phase I Cohort were included in this analysis.
Measure: Mean (Standard Error); unit: percentage fidelity achieved
Arm/Group | LOCI (Intervention) | Training and Technical Assistance Only (Control)
Number analyzed (Participants) | 117 | 117
percentage fidelity achieved | 23.1 (9.0) | 3.4 (2.5)
Statistical Analysis 1: Comparison: LOCI (Intervention) vs Training and Technical Assistance Only (Control); Test type: Superiority; p = .014, Mixed Models Analysis

2. Primary Outcome: Change From Baseline to 6-months in Youth Total Problems Score on the Short Form Assessment for Children (SAC) - Phase I Cohort
Description: The SAC Total Problem Score is a 48-item measure of youth internalizing (e.g., anxious, depressed) and externalizing (e.g., aggressive, noncompliant, overactive) behaviors (range=0-96) completed by caregivers of youth. Total Problem Score was assessed at baseline (youth's entry into treatment) and monthly for 6 months, change from baseline to month 6 is reported.
Time Frame: 0-6 months after youth's baseline/ entry into treatment
Population: Analysis includes youths from Phase I cohort.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | LOCI (Intervention) | Training and Technical Assistance Only (Control)
Number analyzed (Participants) | 117 | 117
units on a scale | -8.17 (1.19) | -4.04 (1.15)
Statistical Analysis 1: Comparison: LOCI (Intervention) vs Training and Technical Assistance Only (Control); Test type: Superiority; p = .023, Mixed Models Analysis

3. Primary Outcome: Percentage Fidelity to the OQ-A System Experienced by the Youth (0-100%)
Description: as for outcome 1
Time Frame: 0-6 months after youth's baseline/ entry into treatment
Population: Analyses based on an intent-to-treat approach. Note that one clinic was identified as an extreme outlier and consequently was excluded from analyses.
Measure: Mean (Standard Error); unit: percentage fidelity achieved
Arm/Group | LOCI (Intervention) | Training and Technical Assistance Only (Control)
Number analyzed (Participants) | 269 | 146
percentage fidelity achieved | 5.65 (4.79) | 0.97 (1.27)
Statistical Analysis 1: Comparison: LOCI (Intervention) vs Training and Technical Assistance Only (Control); Test type: Superiority; p = .188, Mixed Models Analysis

4. Primary Outcome: Change From Baseline to 6-months in Youth Total Problems Score on the Short-form Assessment for Children (SAC) - Phase II Cohort
Description: as for outcome 2
Time Frame: 0-6 months after youth's baseline/ entry into treatment
Population: One clinic was excluded from analyses because it was an extreme outlier.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | LOCI (Intervention) | Training and Technical Assistance Only (Control)
Number analyzed (Participants) | 269 | 146
units on a scale | -4.82 (.70) | -5.19 (1.02)
Statistical Analysis 1: Comparison: LOCI (Intervention) vs Training and Technical Assistance Only (Control); Test type: Superiority; p = .782, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected for caregivers, who were the ones formally enrolled in the study.
Description: Because adverse event data were not collected for caregiver participants, the numbers at risk in each category below equal zero.
Arm/Group | LOCI (Intervention) | Training and Technical Assistance Only (Control)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT04096274/Prot_SAP_000.pdf